CLINICAL TRIAL: NCT03541811
Title: Joint-health Outcome Scoring: Exploration in Patients With Hemophilia in Austria (JOSEPHA Phase 1)
Brief Title: Gait Examination in Patients With Hemophilia in Austria
Acronym: JOSEPHA
Status: Completed | Type: Observational
Sponsor: FH Campus Wien, University of Applied Sciences (Other)
Collaborators: Medical University of Vienna (Other); Shire (Industry)
Responsible Party: Principal Investigator, Peter Putz, Researcher, FH Campus Wien, University of Applied Sciences
Other Study IDs: JOSEPHA Phase 1
Record Dates: First submitted 2018-04-03; First posted 2018-05-31 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Hemophilia
Keywords: gait; motion capture; hemophilia joint health score; physical activity; body composition; gait deviation index; hemophilia
MeSH Terms: conditions — Hemophilia A; Motor Activity | interventions — Environmental Biomarkers; Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood, urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with hemophilia (16-45y): not applicable (no intervention administered)
  Interventions: Diagnostic Test: 3-d gait examination (level walking); Diagnostic Test: Anthropometrics and body composition assessment; Diagnostic Test: Biomarkers; Diagnostic Test: Clinical examination; Diagnostic Test: Habitual physical activity tracking (accelerometer based)
- peer-matched healthy control: not applicable (no intervention administered)
  Interventions: Diagnostic Test: 3-d gait examination (level walking); Diagnostic Test: Anthropometrics and body composition assessment; Diagnostic Test: Biomarkers; Diagnostic Test: Clinical examination; Diagnostic Test: Habitual physical activity tracking (accelerometer based)

INTERVENTIONS:
Diagnostic Test: 3-d gait examination (level walking) — Instrumented 3d-gait-analysis will be carried out in the movement lab of the FH (Fachhochschule; University of Applied Sciences) Campus Wien - University of Applied Sciences. The system used is a 10 camera T40S Vicon system with two floor-mounted AMTI OR6/7-2000 force plates. For assessing gait the Plug-in-Gait Lower Body Model with 14 mm retroreflective skin-mounted markers is implemented in the capturing software Vicon Nexus 2.2. The specific parameters will be extracted from the reporting software Vicon Polygon 4.2.
  Markers will be placed by one experienced examiner. Subjects will be instructed to walk barefoot on a 10 meters walkway at self-paced walking speed until five right and five left valid first force plate strikes are captured.
  Other Names: Vicon
Diagnostic Test: Anthropometrics and body composition assessment — Body height will be measured with the stadiometer Seca 213 to the next 0.1cm. Body size and weight will be measured without shoes and outerwear. A correction of 1 kg will be subtracted for clothing. Body weight and body composition will be assessed with the medical body composition analyzer Seca mBCA 515 based on bioelectric impedance analysis.
Diagnostic Test: Biomarkers — Blood will be collected into Vacuette serum-separating tubes and will be kept at room temperature for 30 min. Samples will be centrifuged at 1500g for 10 min and serum aliquots will be stored at 80 C until use. Urine samples will be collected into Vacuette tubes containing no additive from non-fasted individuals between 8:00 and 12:00 a.m. Urine samples will be kept at 4 °C for a maximum of 8 h, and then aliquoted and stored at 80 °C.
  All biomarkers (except vitamin D and CRP) will be measured in duplicates using standard enzyme-linked immunosorbent assay (ELISA) kits. Serum samples will be assessed for the level of sCOMP, sC1,2C, and sCS846, IL-6, IL-1, sTNFR1 and sTNFR2. Vitamin D and CRP will be measured using automated immunoassay. In urine samples uCTX-II will be determined and these levels will be corrected for creatinine levels (Jaffé method, in-house validated method).
Diagnostic Test: Clinical examination — Hemophilia joint health score (HJHS) will be assessed. Height will be measured with a stadiometer (SECA 213), weight with a medical scale (Marsden M-420) and leg length according to the Plug-in-Gait protocol with a measuring tape from the Anterior Spina Iliaca Superior to the distal aspect of the Medial Malleolus. Further anthropometrical parameters taken will be knee distance and malleoli distance by using a caliper. Gait relevant passive joint ROM of the knee, hip and ankle will be assessed by means of a handheld goniometer. The flexibility of hamstring muscles will be expressed as Popliteal Angle measured with a goniometer with the subjects supine and the hip in 90° flexion.
Diagnostic Test: Habitual physical activity tracking (accelerometer based) — Participants will be instructed to wear an Actigraph wGT3X-BT tri-axial accelerometer permanently over a period of seven consecutive days with an elastic band on right hand sided hip. Data will be process with software ActiLife version 6.13. Cut-offs of at least 10 hours daily wear-time and a minimum of three valid weekdays and one valid weekend day will be applied for data cleaning. Count sampling epoch will be set at one minute. The so called Freedson Adult VM2 Cut-Offs will be applied to categorize physical activity intensities. The so called Freedson VM3 Combination will be applied for the estimation of activity energy expenditure.
  Other Names: ActiGraph GT9X Link

SUMMARY:
Hemophilia is an inherited disease caused by deficiency in varying degrees of clotting factors VIII and IX. Depending on the percentage of clotting factor in the blood the disease is categorized as "severe" (<1%, characterized by spontaneous bleedings), "moderate" (1-5%) and "mild" (>5%). If untreated, recurrent bleeding into the synovial joints often results in irreversible damage due to destruction of the cartilages and progressive joint impairment.

3d-gait analysis has been demonstrated as valid method to assess abnormal gait patterns and to monitor disease progression in patients with hemophilia (PWH). Furthermore, its outcomes facilitate the design of individually tailored therapeutic programs. In contrast to radiological examinations, 3d-gait analyses take place under weight-bearing conditions, which is a relevant issue in terms of weight-induced pain.

This study aims to explore the applicability of 3-d gait analysis as biomarker (gait deviation index) for functional impairments in PWH. Besides 3-d gait scores, secondary endpoints such as biomarkers reflecting cartilage damage and a laterality-ratio of leg muscle mass (in the case of one-sided target joints) will be tested for their ability to detect functional impairments in young adults with hemophilia.

Based on sample size calculation, 24 subjects aged 16-49 years, able to walk without aids or assistance will be included in each of the two groups: control (healthy, male), PWH (severe or moderate, treated prophylactically). Subjects suffering from functional impairments caused by other conditions than hemophilia, patients with bleedings within 30 days prior to the examination, PWH treated with immune-tolerance therapy and/or not successfully treated present or past high-titer factor VIII or FIX inhibitor will be excluded.

Subjects will pass through a set of examinations (medical history, clinical examination, 3d-gait analysis, anthropometrics, body composition analysis, venipuncture, and urine sampling) and carry an accelerometer device for seven consecutive days.

Confounder adjusted group differences will be assessed by ANCOVA with contrasts and Bonferroni correction. Correlations between the applied examination approaches will be assessed.

An evidence based health promotion program including follow-up examinations, physical activity promotion, and tailored physiotherapy are being envisaged as a follow-up project (JOSEPHA phase 2).

ELIGIBILITY:
Inclusion Criteria (test group):

* Provide signed and dated informed consent form (additionally from guardian for participants aged under 18 years)
* Willing to comply with all study procedures and be available for the duration of the study
* Diagnosed severe or moderate hemophilia A or B
* Age between 16 and 49 years
* Able to walk without aids or assistance
* Treated with prophylactic substitution, initiated until the age of 18 years

Inclusion Criteria (control group):

* Provide signed and dated informed consent form (additionally from guardian for participants aged under 18 years)
* Willing to comply with all study procedures and be available for the duration of the study
* Male
* Age between 16 and 49 years (no blood samples for participants aged under 18 years)
* Physiological and symmetric gait pattern without using aids or assistance

Exclusion Criteria:

* Subjects suffering from functional impairments caused by other conditions than hemophilia
* PWH with joint bleedings within 30 days prior to the examination (applies for test group only)
* PWH treated with immune-tolerance therapy and/or not successfully treated present or past high-titer factor VIII or FIX inhibitor (applies for test group only)

Ages: 16 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Test group population will be recruited at the clinical hemophilia center and pediatric unit of the Medical University of Vienna (patients with hemophila have biannual appointments)
  Test group participants are asked to invite a friend at the same age (+/- 3 years; between 16 and 45y) to participate in the sense of a peer-matched control
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Gait Deviation Index (GDI) | May 2018 - Oct 2018 (anticipated)
  Score expressing overall gait physiology; resulting from 3-d gait analysis [dimensionless]

SECONDARY OUTCOMES:
Kinematic gait parameters | May 2018 - Oct 2018 (anticipated)
  Functional range of motion Hip, Knee, Ankle [°]
Walking velocity | May 2018 - Oct 2018 (anticipated)
  [m sec-1]
Walking cadence | May 2018 - Oct 2018 (anticipated)
  [steps min-1]
Step length | May 2018 - Oct 2018 (anticipated)
  [m]
Stance phase duration | May 2018 - Oct 2018 (anticipated)
  [% gait cycle]
Swing phase duration | May 2018 - Oct 2018 (anticipated)
  [% gait cycle]
Body composition analysis | May 2018 - Oct 2018 (anticipated)
  Bioelectrical impedance derived body fat rate [kg, %], fat-free mass [kg, %]
Biomarkers measured from serum and urine | May 2018 - Oct 2018 (anticipated)
  sCOMP, sC1,2C, sCS846, uCTX-II, Vit D, CRP
Background factors (age) | May 2018 - Oct 2018 (anticipated)
  [years]
Background factors (level of education) | May 2018 - Oct 2018 (anticipated)
  International Standard Classification of Education (ISCED)
Background factors (type and severity of hemophilia) | May 2018 - Oct 2018 (anticipated)
  Type and severity of hemophilia
Background factors (type and history of substitutional therapy ) | May 2018 - Oct 2018 (anticipated)
  Type and history of substitutional therapy
Background factors (history of joint bleedings) | May 2018 - Oct 2018 (anticipated)
  annualized bleeding rate
Background factors (inhibitors & immune-tolerance therapy) | May 2018 - Oct 2018 (anticipated)
  Inhibitors & immune-tolerance therapy history
Hemophilia joint health score (HJHS) | May 2018 - Oct 2018 (anticipated)
  Clinical score [dimensionless]

CONTACTS AND LOCATIONS:
Overall Officials: Peter Putz, Dr, Principal Investigator — FH Campus Wien, Department Health Sciences
Locations (1):
- FH Campus Wien - University of Applied Sciences, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No